CLINICAL TRIAL: NCT04747366
Title: National Pandemic Cohort Network - High-resolution Platform (HAP) Analysis of the Pathophysiology and Pathology of Coronavirus Disease 2019 (COVID-19), Including Chronic Morbidity
Brief Title: Analysis of the Pathophysiology and Pathology of Coronavirus Disease 2019 (COVID-19), Including Chronic Morbidity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Network University Medicine NUM (Unknown); Berlin Institute of Health (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Martin Witzenrath, Prof. Dr. med., Charite University, Berlin, Germany
Other Study IDs: NAPKON-HAP
Record Dates: First submitted 2021-01-20; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Covid19
Keywords: COVID-19; coronavirus; SARS-CoV-2; cohort; observational; phenotyping; NAPKON-HAP; NAPKON; chronic morbidity; pa-covid
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — Saliva, Urin, Oropharyngeal / Nasopharyngeal swab / Bronchoalveolar lavage (BAL) / Endotracheal aspirate (ENTA), whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
NAPKON-HAP is the deep phenotyping platform of the National Pandemic Cohort Network (NAPKON) in Germany. NAPKON is a data and biospecimen collection of patients with COVID-19 and is part of the University Medicine Network (NUM) in Germany. The primary objective of the study is to provide a comprehensive collection of data and biosamples for researchers from national consortia and for participation in international research collaborations for studying COVID-19 and future pandemics.

Data is collected from patients with COVID-19 three times per week during their hospitalization and at follow-up visits after hospital discharge 3, 6, 12, 24, and 36 months after symptom onset. Data include epidemiological and demographic parameters, medical history and potential risk factors, documentation of routine medical procedures, and clinical course, including different patterns of organ involvement, quality of care, morbidity, and quality of life. Moreover, extensive serial high-quality bio sampling consisting of various sample types is performed to allow deep molecular, immunological, and virological phenotyping.

Patients not requiring Intensive Care Unit (ICU)/ Intermediate Care (IMC) treatment will receive 7 and patients requiring ICU/IMC treatment will receive 16 full-phenotyping visits including sampling for biobanking. During hospitalisation the planned blood sampling rate in total is 35 ml at each visit. The total amounts and/or sampling dates may differ according to the ethics committee's regulations for different study centers.

At follow-up visits, the clinical assessment includes an update of the medical history and recent medical events from which additional clinical data is collected (i.e. outpatient CT-scans, echocardiography, external laboratory data). Clinical symptoms are recorded and a physical examination will be performed. Vital signs are recorded and routine blood testing and biosampling is continued. Quality of life is measured with patient-reported outcome questionnaires.

Follow-up visits at months 3 and 12 are "deep phenotyping" visits with a comprehensive and detailed set of examinations. In the following visits at months 24 and 36, only examinations with pathologic results from the last deep phenotyping visit at month 12 will be performed.

A shorter follow-up visit to record quality of life, recent medical events and with a reduced number of examinations focusing on cardiorespiratory performance will take place at month 6.

In case of relevant medical events, new medical information or changes in the participant´s health status, an unscheduled visit can take place anytime within the entire study period.

Data collection during follow up includes standardized quality of life assessment including PROMIS® (Patient-Reported Outcomes Measurement Information System). The pulmonary characterization will include body plethysmography, diffusion capacity, respiratory muscles strength measurement, spiroergometry, capillary blood gas analysis and lung imaging studies (low-dose Computed Tomography (CT), Magnetic Resonance Imaging (MRI) of the lung). Cardiological phenotyping includes echocardiography, electrocardiogram (ECG), 24h-ECG, 24h-blood pressure monitoring, stress cardiac MRI and pulse wave analysis. Neurocognitive testing includes brain MRI, electroencephalogram (EEG), somatosensory testing, refractometry (Visit 3 and 12 months), physical activity test, neurocognitive tests, somatosensory phenotyping, taste- and smell-test. Endocrinological phenotyping will incorporate Advanced Glycation Endproducts (AGE) reader, continuous glucose monitoring for 14 days, Air Displacement Plethysmography (ADP) or bioelectrical impedance analysis (BIA).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Willingness to participate in the study (consent to participate by patient or appropriate legal representative) or inclusion via deferred consent
* Hospitalization at time of enrollment
* Positive evidence for SARS-CoV-2 infection with PCR (polymerase chain reaction) or initial positive rapid diagnostic test in conjunction with typical clinical symptoms, confirmed by a later positive PCR test.

Exclusion Criteria:

* Refusal to participate by patient, or appropriate legal representative
* Any condition that prohibits supplemental blood-sampling beyond routine blood drawing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients, hospitalised at any of the participating hospitals (see study sites) over the age of 18 years, who are willing and deemed able to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2020-11-06 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Patient-reported Quality of life recorded with the help of the European Quality of Life 5 Dimensions 5 Level Version (Eq5d5l) questionnaire | day 1 of enrollment in the study, immediately before discharge, 3, 12, 24 and 36 months after symptom onset
  Health related quality of life after hospital discharge will be assessed with the questionnaire European Quality of Life 5 Dimensions 5 Level Version (Eq5d5l)
Changes in Patient-reported Quality of life recorded with the help of the Short Form Health 36 (Sf36) | day 1 of enrollment in the study, immediately before discharge, 3, 12, 24 and 36 months after symptom onset
  Health related quality of life after hospital discharge will be assessed with the questionnaire Short Form Health 36 (Sf36)
Changes in Patient-reported Quality of life recorded with the help of the Patient-Reported Outcomes Measurement Information System (PROMIS Profile) | day 1 of enrollment in the study, immediately before discharge, 3, 12, 24 and 36 months after symptom onset
  Health related quality of life after hospital discharge will be assessed with the questionnaire Patient-Reported Outcomes Measurement Information System (PROMIS Profile)
Changes in Patient-reported Quality of life recorded with the help of the Neuropathy Questionnaire (Mnsi) | day 1 of enrollment in the study, immediately before discharge, 3, 12, 24 and 36 months after symptom onset
  Health related quality of life after hospital discharge will be assessed with the questionnaire Neuropathy Questionnaire (Mnsi)
Changes in Patient-reported Quality of life recorded with the help of the Trauma Patient Health Questionnaire | day 1 of enrollment in the study, immediately before discharge, 3, 12, 24 and 36 months after symptom onset
  Health related quality of life after hospital discharge will be assessed with the questionnaire Trauma Patient Health Questionnaire
Changes in Patient-reported Quality of life recorded with the help of the PTSD (Post-traumatic stress disorder) Checklist for Diagnostic and Statistical Manual of Mental Disorders 5 (PCL-5). | day 1 of enrollment in the study, immediately before discharge, 3, 12, 24 and 36 months after symptom onset
  Health related quality of life after hospital discharge will be assessed with the PTSD (Post-traumatic stress disorder) Checklist for Diagnostic and Statistical Manual of Mental Disorders 5 (PCL-5). The PTSD Checklist for DSM-5 is a 20-questions self-report measure that assesses the presence and severity of PTSD symptoms.
Changes in Patient-reported Quality of life recorded with the help of the National Eye Institute Visual Function Questionnaire (NEI-VFQ) | day 1 of enrollment in the study, immediately before discharge, 3, 12, 24 and 36 months after symptom onset
  Health related quality of life after hospital discharge will be assessed with the questionnaire National Eye Institute Visual Function Questionnaire (NEI-VFQ)
Changes in Patient-reported Quality of life recorded with the help of the St. George's Respiratory Questionnaire (SGRQ) | day 1 of enrollment in the study, immediately before discharge, 3, 12, 24 and 36 months after symptom onset
  Health related quality of life after hospital discharge will be assessed with the questionnaire St. George's Respiratory Questionnaire (SGRQ)
Changes in neruocognitive testing with Cambridge Neuropsychological Test Automated Battery (CANTAB) | at follow-up visits (3 and 12 months after symptom onset and 24 and 36 months after symptom onset (only in case of abnormal results)
  CANTAB tests can detect changes in neuropsychological performance and include tests of working memory, learning and executive function; visual, verbal and episodic memory; attention, information processing and reaction time; social and emotion recognition, decision making and response control.
Changes in neruocognitive testing with Montreal Cognitive Assessment Test (MOCA) | at follow-up visits (3 and 12 months after symptom onset and 24 and 36 months after symptom onset (only in case of abnormal results)
  This test is a screening procedure to determine cognitive deficits. Central cognitive functions are examined using 11 task complexes. This includes time and spatial orientation, learning and memory, attention, language and language skills, reading, writing, drawing and calculating (test duration approx. 10 minutes).
Changes in blood pressure measured during spiroergometry testing | at follow-up visits (3 and 12 months after symptom onset and 24 and 36 months after symptom onset (only in case of abnormal results)
  Spiroergometry (spirometry while the participant exercises on a bicycle ergometer) is used to evaluate physical performance and fitness. Using spiroergometry blood pressure is measured during the test and compared with normative values.
Changes in sensomotory testing with the questionnaire for peripheral neuropathy (Michigan Neuropathy Screening Instrument, MNSI) | at follow-up visits (3 and 12 months after symptom onset and 24 and 36 months after symptom onset (only in case of abnormal results)
  The MNSI will be used to screen patients for peripheral neuropathy.
Changes in sensomotory testing with the questionnaire (painDETECT-questionnaire, pDQ) | at follow-up visits (3 and 12 months after symptom onset and 24 and 36 months after symptom onset (only in case of abnormal results)
  PainDETECT will be used to screen patients for for neuropathic pain.
Changes in Quantitative sensory testing (QST) | at follow-up visits (3 and 12 months after symptom onset and 24 and 36 months after symptom onset (only in case of abnormal results)
  Quantitative sensory testing (QST) is a method for semiquantative evaluation of somatosensory nervous system disorders, including chronic pain and pain related to various diseases. It essentially determines the sensation and pain thresholds for cold and warm temperatures, and the vibration sensation threshold by stimulating the skin and comparing the results to normative values.
Changes in Point-of-care neurography | at follow-up visits (3 and 12 months after symptom onset and 24 and 36 months after symptom onset (only in case of abnormal results)
  Point-of-care neuography measures nerve conduction using a point-of-care device (DPNcheck, Neurometrix Inc, USA).
Changes in pulmonary function assessed by body plethysmography | immediately before discharge, at follow-up visits (3, 6 and 12 months after symptom onset and 24 and 36 months after symptom onset (only in case of abnormal results)
  Body plethysmography will yield information on the static and dynamic lung volumes to assess obstructive and restrictive ventilation patterns.
Changes in pulmonary function assessed by single breath CO (carbon monoxide) diffusion capacity (DLCO) | immediately before discharge, at follow-up visits (3, 6 and 12 months after symptom onset and 24 and 36 months after symptom onset (only in case of abnormal results)
  The DLCO test provides a general assessment of the lungs' ability to take up oxygen from the inspiratory air and to release carbon dioxide.
Changes in heart rate measured with ECG (Electrocardiogram) during spiroergometry testing | at follow-up visits (3 and 12 months after symptom onset and 24 and 36 months after symptom onset (only in case of abnormal results)
  Spiroergometry (spirometry while the participant exercises on a bicycle ergometer) is used to evaluate physical performance and fitness. ECG is a test, used to monitor the electrical activity of the heart. Standard placement of 12-lead electrodes will be used. The patient´s heart rate will be assessed longitudinally and compared to normative values.
Changes in the oxygen saturation of the blood measured during spiroergometry testing | at follow-up visits (3 and 12 months after symptom onset and 24 and 36 months after symptom onset (only in case of abnormal results)
  Spiroergometry (spirometry while the participant exercises on a bicycle ergometer) is used to evaluate physical performance and fitness. Two blood samples are taken 2 hours apart. The first one is taken before the spiroergometry test and the second one - 120 minutes after the first one. The total concentration of carbon dioxide (ctCO2) of the blood is measured and compared with normative values.
Changes in the total concentration of carbon dioxide (ctCO2) of the blood measured during spiroergometry testing | at follow-up visits (3 and 12 months after symptom onset and 24 and 36 months after symptom onset (only in case of abnormal results)
  Spiroergometry (spirometry while the participant exercises on a bicycle ergometer) is used to evaluate physical performance and fitness. The carbon dioxide content of the blood is measured during the test and compared with normative values.
Changes in the pH value of the blood measured during spiroergometry testing | at follow-up visits (3 and 12 months after symptom onset and 24 and 36 months after symptom onset (only in case of abnormal results)
  Spiroergometry (spirometry while the participant exercises on a bicycle ergometer) is used to evaluate physical performance and fitness. Two blood samples are taken 2 hours apart. The first one is taken before the spiroergometry test and the second one - 120 minutes after the first one. The pH value of the blood is measured and compared with normative values. The pH value describes how acidic or basic the blood is.
Changes in the bicarbonate content of the blood measured during spiroergometry testing | at follow-up visits (3 and 12 months after symptom onset and 24 and 36 months after symptom onset (only in case of abnormal results)
  Spiroergometry (spirometry while the participant exercises on a bicycle ergometer) is used to evaluate physical performance and fitness. Two blood samples are taken 2 hours apart. The first one is taken before the spiroergometry test and the second one - 120 minutes after the first one. The bicarbonate content of the blood is measured and compared with normative values. Bicarbonate is a form of carbon dioxide.
Changes in the blood lactate levels during spiroergometry testing | at follow-up visits (3 and 12 months after symptom onset and 24 and 36 months after symptom onset (only in case of abnormal results)
  Spiroergometry (spirometry while the participant exercises on a bicycle ergometer) is used to evaluate physical performance and fitness. Two blood samples are taken 2 hours apart. The first one is taken before the spiroergometry test and the second one - 120 minutes after the first one. The lactate saturation is measured and compared with normative values.
Changes in the partial pressure of carbon dioxide (pCO2) of the blood measured during spiroergometry testing | at follow-up visits (3 and 12 months after symptom onset and 24 and 36 months after symptom onset (only in case of abnormal results)
  Spiroergometry (spirometry while the participant exercises on a bicycle ergometer) is used to evaluate physical performance and fitness. Two blood samples are taken 2 hours apart. The first one is taken before the spiroergometry test and the second one - 120 minutes after the first one. The partial pressure of carbon dioxide (pCO2) of the blood is measured and compared with normative values.
Changes in heart rhythm type measured with ECG (Electrocardiogram) during spiroergometry testing | at follow-up visits (3 and 12 months after symptom onset and 24 and 36 months after symptom onset (only in case of abnormal results
  Spiroergometry (spirometry while the participant exercises on a bicycle ergometer) is used to evaluate physical performance and fitness. ECG is a test, used to monitor the electrical activity of the heart. Standard placement of 12-lead electrodes will be used. The patient´s heart rhythm will be assessed. Any abnormalities (too slow, too fast, irregular) will be documented and subsequently clinical consequences are being taken.
Changes in time intervals of PQ measured with ECG (Electrocardiogram) during spiroergometry testing | at follow-up visits (3 and 12 months after symptom onset and 24 and 36 months after symptom onset (only in case of abnormal results)
  Spiroergometry (spirometry while the participant exercises on a bicycle ergometer) is used to evaluate physical performance and fitness. ECG is a test, used to monitor the electrical activity of the heart. Standard placement of 12-lead electrodes will be used. The time interval of PQ corresponds to the time interval from the beginning of the P wave to the beginning of the Q wave of the QRS complex. The time interval of PQ gives us information about the time required for the action potential to be transmitted from the atria to the ventricles. The recorded PQ time will be compared to normative values. In case of delayed PQ times, further diagnostic is carried out according to current guidelines.
Changes in time intervals of QRS measured with ECG (Electrocardiogram) during spiroergometry testing | at follow-up visits (3 and 12 months after symptom onset and 24 and 36 months after symptom onset (only in case of abnormal results)
  Spiroergometry (spirometry while the participant exercises on a bicycle ergometer) is used to evaluate physical performance and fitness. ECG is a test, used to monitor the electrical activity of the heart. Standard placement of 12-lead electrodes will be used. The QRS complex is combination of the Q wave, R wave and S wave. The time interval of QRS corresponds to the time needed for ventricular depolarization. The recorded QRS time will be compared to normative values. In case of new diagnosed bundle blocks, further diagnostic is carried out according to current guidelines.
Changes in time intervals of QT measured with ECG (Electrocardiogram) during spiroergometry testing | at follow-up visits (3 and 12 months after symptom onset and 24 and 36 months after symptom onset (only in case of abnormal results)
  Spiroergometry (spirometry while the participant exercises on a bicycle ergometer) is used to evaluate physical performance and fitness. ECG is a test, used to monitor the electrical activity of the heart. Standard placement of 12-lead electrodes will be used. The time interval of QT corresponds to the time interval from the beginning of the Q wave to the end of the T wave. The time interval of QT gives us information about the time required for ventricular depolarisation and repolarisation. The recorded QT time will be compared to normative values. In case of abnormal QT times, further diagnostic is carried out according to current guidelines.
Deviations in the ST segment depicted with the use of ECG (Electrocardiogram) during spiroergometry testing | at follow-up visits (3 and 12 months after symptom onset and 24 and 36 months after symptom onset (only in case of abnormal results)
  Spiroergometry (spirometry while the participant exercises on a bicycle ergometer) is used to evaluate physical performance and fitness. ECG is a test, used to monitor the electrical activity of the heart. Standard placement of 12-lead electrodes will be used. The ST-segment is a section between the end of the S wave and the beginning of the T wave and reflects the depolarized state and initial repolarization of the ventricles. Deviations in the ST segment (elevation or depression) will be documented. In case of ST segment elevation or depression, further diagnostic is carried out according to current guidelines.

SECONDARY OUTCOMES:
Changes in body temperature | every day during hospitalisation (from date of admission in trial until date of discharge or date of death, assessed up to 100 weeks
  Assessment of the patient´s body temperature will be performed at all visits during the acute phase.
Changes in blood pressure | every day during hospitalisation (from date of admission in trial until date of discharge or date of death, assessed up to 100 weeks
  Assessment of the patient´s blood pressure will be performed at all visits during the acute phase.
Changes in heart rate | every day during hospitalisation (from date of admission in trial until date of discharge or date of death, assessed up to 100 weeks
  Assessment of the patient´s heart rate will be performed at all visits during the acute phase.
Changes in breath frequency (respiratory rate) | every day during hospitalisation (from date of admission in trial until date of discharge or date of death, assessed up to 100 weeks
  Assessment of the patient´s breath frequency (respiratory rate) will be performed at all visits during the acute phase.
Changes in peripheral oxygen saturation | every day during hospitalisation (from date of admission in trial until date of discharge or date of death, assessed up to 100 weeks
  Assessment of the patient´s peripheral oxygen saturation will be performed at all visits during the acute phase.
Changes in the clinical score SOFA (sequential organ failure assessment) | at primary admission to hospital, upon admission to ICU ward, every Monday, Wednesday and Friday during ICU ward stay, assessed up to 100 weeks
  At each study visit on the ICU ward, the SOFA score will be assessed (if provided in the clinical information system).
Changes in the clinical score Berlin ARDS (acute respiratory distress syndrome) severity score (if provided) | every Monday, Wednesday and Friday during ICU ward stay, assessed up to 100 weeks
  At each study visit on the ICU ward, the Berlin ARDS (acute respiratory distress syndrome) severity score will be assessed (if provided in the clinical information system).
Changes in the clinical score APACHE (Acute Physiology and Chronic Health Evaluation) Score | upon admission to ICU
  At each study visit on the ICU ward, the APACHE (Acute Physiology and Chronic Health Evaluation) score will be assessed (if provided in the clinical information system).
Changes in the clinical score NEWS (National Early Warning Score) | day 1 of enrollment in the study (day of hospitalization), if available
  At primary admission to hospital NEWS (National Early Warning Score) will be assessed (if provided in the clinical information system).
Changes in the clinical score qSOFA Score (quick sequential organ failure assessment) | day 1 of enrollment in the study (day of hospitalization), if available
  At primary admission to hospital qSOFA Score will be assessed (if provided in the clinical information system).
Changes in the Barthel Index | day 1 of enrollment in the study, every Monday, Wednesday and Friday during hospitalisation, (assessed up to 100 weeks?), immediately before discharge, at follow up visits 3, 12, 24 and 36 months after symptom onset
  The changes in the Barthel Index score will be recorded and evaluated, if provided.
Changes in the Frailty score | day 1 of enrollment in the study, every Monday, Wednesday and Friday during hospitalisation, (assessed up to 100 weeks?), immediately before discharge, at follow up visits 3, 12, 24 and 36 months after symptom onset
  At each study visit during hospitalization (visits are conducted 3 times a week until discharge) the Frailty score will be assessed (if provided in the clinical information system).
Changes in the clinical score Murray Score | every Monday, Wednesday and Friday during ICU ward stay, assessed up to 100 weeks
  At each study visit on ICU ward the Murray Score will be assessed (if provided in the clinical information system).
Changes in the clinical score Glasgow Coma Scale (GCS) | upon admission to ICU ward, every Monday, Wednesday and Friday ICU ward stay, assessed up to 100 weeks
  At each study visit on ICU ward the Glasgow Coma Scale score will be assessed (if provided in the clinical information system).
Changes in the clinical score RASS (Richmond Agitation Sedation Scale) | upon admission to ICU ward, every Monday, Wednesday and Friday ICU ward stay, assessed up to 100 weeks
  At each study visit on ICU ward the RASS (Richmond Agitation Sedation Scale)will be assessed (if provided in the clinical information system).
Changes in the clinical score CAM-ICU (Score Confusion Assessment Method for Intensive Care Unit) | every Monday, Wednesday and Friday during ICU ward stay,assessed up to 100 weeks
  At each study visit on ICU ward the CAM-ICU (Score Confusion Assessment Method for Intensive Care Unit) score will be assessed (if provided in the clinical information system).
Changes in the clinical score SAPSII (Simplified acute physiology Score II) | every Monday, Wednesday and Friday during ICU ward stay, assessed up to 100 weeks
  At each study visit on ICU ward the SAPSII (Simplified acute physiology Score II) will be assessed (if provided in the clinical information system).
Changes in the clinical score NRS (numeric rating scale) pain score | every Monday, Wednesday and Friday during ICU ward stay, assessed up to 100 weeks
  At each study visit on ICU ward the NRS (numeric rating scale) pain score will be assessed (if provided in the clinical information system).
Changes in the clinical score BPS (behavioural pain scale) pain score | every Monday, Wednesday and Friday during ICU ward stay, assessed up to 100 weeks
  At each study visit on ICU ward the BPS (behavioural pain scale) pain score will be assessed (if provided in the clinical information system).
Changes in the clinical score CPOT (Critical Care Pain Observation tool) | every Monday, Wednesday and Friday during ICU ward stay, assessed up to 100 weeks
  At each study visit on ICU ward the CPOT (Critical Care Pain Observation tool) score will be assessed (if provided in the clinical information system).
Changes in the clinical score DDS (Delirium detection score) | every Monday, Wednesday and Friday during ICU ward stay, assessed up to 100 weeks
  At each study visit on ICU ward the DDS (Delirium detection score) will be assessed (if provided in the clinical information system).
Changes in the checked items on the ICDSC (Intensive Care Delirium Screening checklist) | every Monday, Wednesday and Friday during ICU ward stay, assessed up to 100 weeks
  At each study visit on ICU ward the ICDSC (Intensive Care Delirium Screening checklist) will be assessed (if provided in the clinical information system).
Changes in the heart time volume | every Monday, Wednesday and Friday during ICU ward stay, assessed up to 100 weeks
  Assessment of the patient´s heart time volume will be performed at all visits during their stay in the ICU ward.
Changes in the cardiac index | every Monday, Wednesday and Friday during ICU ward stay, assessed up to 100 weeks
  Assessment of the patient´s cardiac index will be performed at all visits during their stay in the ICU ward.
Changes in EVLWI (Extravascular Lung Water Index) | every Monday, Wednesday and Friday during ICU ward stay, assessed up to 100 weeks
  Assessment of the patient´s Extravascular Lung Water Index measurement will be performed at all visits during their stay in the ICU ward.
Changes in Systemic Vascular Resistance Index (SVRI) | every Monday, Wednesday and Friday during ICU ward stay, assessed up to 100 weeks
  Assessment of the patient´s Systemic Vascular Resistance Index (SVRI) measurement will be performed at all visits during their stay in the ICU ward.
Changes in ITBVI (Intrathoracic Blood Volume Index) | every Monday, Wednesday and Friday during ICU ward stay, assessed up to 100 weeks
  Assessment of the patient´s ITBVI (Intrathoracic Blood Volume Index) measurement will be performed at all visits during their stay in the ICU ward.
Changes in the score WHO (World Health Organisation) clinical ordinal scale | every day during hospital stay (from day of admission until discharge from hospital, assessed up to 100 weeks) and at follow-up visits (3, 12, 24 and 36 months after symptom onset)
  Changes in the patient´s score on the WHO clinical ordinal scale, used to measure illness severity over time will be assessed.
Changes in the NYHA (New York Heart Association) score | at deep phenotyping during follow-up visits (3 and 12 months after symptom onset)
  The changes in the NYHA (New York Heart Association) score will be recorded and evaluated, if provided.
Changes in the Post-COVID-19 Functional Status (PCFS) scale | at follow-up visits (3, 12, 24 and 36 months after symptom onset)
  The changes in the Post-COVID-19 Functional Status (PCFS) scale will be recorded and evaluated, if provided.
Changes in the National Institutes of Health Stroke Scale (NIHSS) | at deep phenotyping during follow-up visits (3 and 12 months after symptom onset)
  The changes in the National Institutes of Health Stroke Scale (NIHSS) will be recorded and evaluated, if provided.
Changes in the Katz Index | at follow-up visits (3, 12, 24 and 36 months after symptom onset)
  The changes in the Katz Index will be recorded and evaluated, if provided.
Changes in the Rose Dyspnea Scale | at deep phenotyping during follow-up visits (3 and 12 months after symptom onset)
  The changes in the Rose Dyspnea Scale will be recorded and evaluated, if provided.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Witzenrath, Prof. Dr. med., Principal Investigator — Charite University Hospital Berlin
Locations (11):
- Germany (11):
  - University Medical Center Freiburg Department of Internal Medicine II Department of Infectiology, Freiburg im Breisgau, Baden-Wurttemberg
  - University Hospital Heidelberg Clinic for Gastroenterology, Infections, Poisoning, Heidelberg, Baden-Wurttemberg
  - Clinic of the University of Munich Medical Clinic and Polyclinic III, Munich, Bavaria
  - University Hospital Frankfurt Medical Clinic II Department of infectiology, Frankfurt am Main, Hesse
  - University Hospital Giessen (+Marburg) Medical Clinic II Pneumology and internal intensive care medicine Infectiology, Gastroenterology, Nephrology, Giessen, Hesse
  - Hanover Medical School Clinic for Pneumology, Hanover, Lower Saxony
  - University Hospital Cologne Internal Medicine I and Hematology and Oncology, Infectiology, additional qualification in Emergency Medicine, Cologne, North Rhine-Westphalia
  - University Medical Center Schleswig-Holstein (Campus Kiel): Internal medicine, gastroenterology, pneumology, allergology, sleep medicine, emergency medicine, intensive care, Kiel, Schleswig-Holstein
  - University Medical Center Schleswig-Holstein (Campus Lübeck): Internal medicine, gastroenterology, pneumology, allergology, sleep medicine, emergency medicine, intensive care, Lübeck, Schleswig-Holstein
  - University Hospital Jena Department of Internal Medicine IV, Jena, Thuringia
  - Charité University Hospital Berlin Medical Clinic Infectiology and Pneumology CCM/CVK, Berlin

IPD SHARING:
Plan to Share IPD: No
Given a concrete inquiry and prior consent by the study participants in question, IPD (individual participant data) can be made available on a case by case basis.

REFERENCES:
- [Derived] Hartung TJ, Steigerwald F, Romanello A, Kodde C, Endres M, Frank S, Heuschmann P, Koehler P, Krohn S, Pape D, Schaller J, Stocklein S, Vadasz I, Vehreschild J, Witzenrath M, Zoller T, Finke C; NAPKON Study Group. Post-COVID Fatigue Is Associated With Reduced Cortical Thickness After Hospitalization. Ann Clin Transl Neurol. 2025 Nov 25. doi: 10.1002/acn3.70260. Online ahead of print. PMID 41288256
- [Derived] Appel KS, Lee CH, Nunes de Miranda SM, Maier D, Reese JP, Anton G, Bahmer T, Ballhausen S, Balzuweit B, Bellinghausen C, Blumentritt A, Brechtel M, Chaplinskaya-Sobol I, Erber J, Fiedler K, Geisler R, Heyder R, Illig T, Kohls M, Kollek J, Krist L, Lorbeer R, Miljukov O, Mitrov L, Nurnberger C, Pape C, Pley C, Schafer C, Schaller J, Schattschneider M, Scherer M, Schulze N, Stahl D, Stubbe HC, Tamminga T, Tebbe JJ, Vehreschild MJGT, Wiedmann S, Vehreschild JJ. A precise performance-based reimbursement model for the multi-centre NAPKON cohorts - development and evaluation. Sci Rep. 2024 Jun 13;14(1):13607. doi: 10.1038/s41598-024-63945-5. PMID 38871878
- [Derived] Schons M, Pilgram L, Reese JP, Stecher M, Anton G, Appel KS, Bahmer T, Bartschke A, Bellinghausen C, Bernemann I, Brechtel M, Brinkmann F, Brunn C, Dhillon C, Fiessler C, Geisler R, Hamelmann E, Hansch S, Hanses F, Hanss S, Herold S, Heyder R, Hofmann AL, Hopff SM, Horn A, Jakob C, Jiru-Hillmann S, Keil T, Khodamoradi Y, Kohls M, Kraus M, Krefting D, Kunze S, Kurth F, Lieb W, Lippert LJ, Lorbeer R, Lorenz-Depiereux B, Maetzler C, Miljukov O, Nauck M, Pape D, Puntmann V, Reinke L, Rommele C, Rudolph S, Sass J, Schafer C, Schaller J, Schattschneider M, Scheer C, Scherer M, Schmidt S, Schmidt J, Seibel K, Stahl D, Steinbeis F, Stork S, Tauchert M, Tebbe JJ, Thibeault C, Toepfner N, Ungethum K, Vadasz I, Valentin H, Wiedmann S, Zoller T, Nagel E, Krawczak M, von Kalle C, Illig T, Schreiber S, Witzenrath M, Heuschmann P, Vehreschild JJ; NAPKON Research Group. The German National Pandemic Cohort Network (NAPKON): rationale, study design and baseline characteristics. Eur J Epidemiol. 2022 Aug;37(8):849-870. doi: 10.1007/s10654-022-00896-z. Epub 2022 Jul 29. PMID 35904671